CLINICAL TRIAL: NCT01249612
Title: No Effect of Knee Joint Icing on Knee-extension Strength After Total Knee Arthroplasty. A Randomized Cross-over Study
Brief Title: Knee Joint Icing and Knee-extension Strength
Acronym: IS
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Lundbeck Foundation (Other)
Responsible Party: Principal Investigator, Bente Holm, MSc PT, Hvidovre University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: (H-A-2008-063, nr. 24100; TKA-BH3 (Registry Identifier: H-A-2008-063)
Record Dates: First submitted 2010-11-23; First posted 2010-11-30 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: Arthroplasty
Keywords: Knee joint icing; knee-extension strength
MeSH Terms: interventions — Hyperthermia, Induced; Cryotherapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control treatment (Placebo Comparator): Elbow joint icing using two plastic bags with crushed ice
  Interventions: Other: Thermotherapy
- Active treatment (Active Comparator): Knee joint icing using two plastic bags with crushed ice
  Interventions: Other: Thermotherapy

INTERVENTIONS:
Other: Thermotherapy — Knee joint icing
  Other Names: Cryotherapy
  Arms: Active treatment
Other: Thermotherapy — Elbow joint icing
  Other Names: Cryotherapy
  Arms: Control treatment

SUMMARY:
With this study the investigators wish to (1) investigate the acute effect of knee joint icing on knee-extension strength shortly after total knee arthroplasty (TKA); and (2) investigate the acute effect of knee joint icing on knee pain, knee joint circumference and functional performance shortly after TKA.

DETAILED DESCRIPTION:
As knee joint icing had no acute effect on knee-extension strength in the present study, prolonged icing may have an effect on one or more of the parameters, and further studies are needed to determine the potential beneficial effects of cooling after TKA.

ELIGIBILITY:
Inclusion Criteria:

* primary unilateral total knee arthroplasty

Exclusion Criteria:

* inability to speak and understand Danish
* inability to perform the measurements due to other diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-04; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Knee-extension strength | In the first week after surgery patients are measured on two days: One day before and after active (knee icing) treatment and one day before and after control (elbow icing) treatment
  Maximal knee-extension strength is measured using a hand-held dynamometer

SECONDARY OUTCOMES:
Knee pain | In the first week after surgery patients are measured on two days: One day before and after active (knee icing) treatment and one day before and after control (elbow icing) treatment
  Knee pain was quantified by using The Visual Analog Scale (VAS) at rest and during active measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Bente Holm, MSc, Principal Investigator — Department of Orthopaedic Surgery, University Hospital at Hvidovre, Kettegaard Alle 30, DK-2650 Hvidovre, Denmark
Locations (1):
- The Lundbeckcenter for fast-track hip and knee surgery, Copenhagen, Hvidovre, Denmark

REFERENCES:
- [Derived] Holm B, Husted H, Kehlet H, Bandholm T. Effect of knee joint icing on knee extension strength and knee pain early after total knee arthroplasty: a randomized cross-over study. Clin Rehabil. 2012 Aug;26(8):716-23. doi: 10.1177/0269215511432017. Epub 2012 Jan 19. PMID 22261815